CLINICAL TRIAL: NCT00957268
Title: A Comparative, Randomized, Open-Label, Multi-Center, Single Dose Pharmacokinetic, Pharmacodynamic and Safety Study of Alogliptin (12.5 mg and 25 mg) Between Children, Adolescents, and Adults With Type 2 (Non-Insulin Dependent) Diabetes Mellitus
Brief Title: Pharmacokinetics, Pharmacodynamics, and Safety of Alogliptin in Children, Adolescents and Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SYR-322_104; 2009-011221-13 (Registry Identifier: EudraCT); U1111-1111-7810 (Registry Identifier: WHO)
Record Dates: First submitted 2009-08-06; First posted 2009-08-12 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Non-insulin dependent diabetes mellitus; Drug therapy; Pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Alogliptin 12.5 mg (age 10 to < 14 years) (Experimental): Alogliptin 12.5 mg, tablets, orally, 1 dose only.
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg (age 10 to < 14 years) (Experimental): Alogliptin 25 mg, tablets, orally, 1 dose only.
  Interventions: Drug: Alogliptin
- Alogliptin 12.5 mg (age 14 to < 18 years) (Experimental): Alogliptin 12.5 mg, tablets, orally, 1 dose only.
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg (age 14 to < 18 years) (Experimental): Alogliptin 25 mg, tablets, orally, 1 dose only.
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg (age 18 to 65 years) (Experimental): Alogliptin 25 mg, tablets, orally, 1 dose only.
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: SYR-322

SUMMARY:
The purpose of this study is to determine the pharmacokinetic and safety profile of alogliptin in children, adolescents, and adults with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Alogliptin is a selective, orally available inhibitor of dipeptidyl peptidase-4 being developed by Takeda Global Research & Development as a treatment for type 2 diabetes mellitus. Inhibition of dipeptidyl peptidase-4 (DPP-4) prolongs the action of 2 important incretin hormones, glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP). These hormones are responsible for increasing insulin synthesis, regulating β-cell proliferation, inhibiting gastric emptying, and inhibiting glucagon secretion.

To date, alogliptin has not been studied in participants less than 18 years of age. As with adults, there is growing evidence of an increase in the prevalence of type 2 diabetes mellitus in children and adolescents.

This study is designed to determine the pharmacokinetic, pharmacodynamic, and safety profiles of alogliptin in children and adolescents with type 2 diabetes mellitus. These profiles will be compared with those of similarly matched adult participants with type 2 diabetes mellitus. Pharmacokinetic, pharmacodynamics, and safety endpoints will be analyzed.

ELIGIBILITY:
Inclusion criteria for children and adolescent participants only (Groups 1 and 2, respectively):

1. Participant was male or female between 10 and 17 years of age.
2. Participant or parent or legal guardian was capable of understanding and complying with the protocol requirements.
3. Participant was capable of understanding an informed consent form (ICF) or assenting to participate. The parent or legal guardian of the participant must have been able to understand and sign an ICF prior to the initiation of any study procedures.
4. Participant weighed at least 36 kg (79 pounds) and had a Screening body mass index (BMI) of at least 18 kg/m^2.
5. Participants had a diagnosis of type 2 diabetes mellitus (T2DM) (non-insulin dependent) based on diagnostic criteria of the American Diabetes Association (ADA). Criteria included:

   1. Fasting plasma glucose level of ≥ 126 mg/dL where fasting is defined as no caloric intake for at least 8 hours, or
   2. 2-hour plasma glucose level of ≥ 200 mg/dL during an oral glucose tolerance test, or
   3. random plasma glucose level of ≥ 200 mg/dL, or
   4. glycated hemoglobin (HbA1c) ≥ 6.5%.
6. Diagnosis could have been historical (documented), or participants could have been diagnosed for this study.
7. Participants had a fasting serum C-peptide concentration ≥ 0.8 ng/mL (≥ 0.26 nmol/L) at the Screening Visit only.
8. Participants may have been taking concomitant metformin if the dose was stable for at least 30 days prior to Day 1 (day of first dosing).

   Inclusion criteria for adult participants only (Group 3):
9. Participant was male or female, and between 18 and 65 years of age, inclusive for gender and race matched adult participants with T2DM only.
10. Participant was capable of understanding and complying with protocol requirements and was willing to sign the ICF prior to the initiation of any study procedures for gender and race matched adult participants with T2DM only.
11. Participant weighed at least 50 kg (110 pounds) and had a Screening BMI between 23 kg/m^2 and 45 kg/m^2 (except for Asian or Asian-descendant participants for whom the range was between 20 kg/m^2 and 35 kg/m^2), inclusive for gender and race matched T2DM adult participants only.
12. Participants had a diagnosis of T2DM (non-insulin dependent) based on diagnostic criteria of the ADA. Criteria included:

    1. Fasting plasma glucose level of ≥ 126 mg/dL where fasting is defined as no caloric intake for at least 8 hours, or
    2. 2-hour plasma glucose level of ≥ 200 mg/dL during an oral glucose tolerance test, or
    3. random plasma glucose level of ≥ 200 mg/dL, or
    4. HbA1c ≥ 6.5%.
13. Diagnosis could have been historical (documented) or participants could have been diagnosed for this study.
14. Participants may have been taking concomitant metformin if the dose was stable for at least 30 days prior to Day 1.
15. Participants may have been taking statin or antihypertensive drugs if the dose was stable for at least 30 days prior to Day 1.

    Inclusion criteria for all participants (Groups 1, 2, and 3):
16. Female participants of childbearing potential and male participants who were sexually active agreed to routinely use adequate contraception from Screening until 30 days after receiving the dose of study drug. NOTE: Women not of childbearing potential were defined as those who were surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation) or who were postmenopausal (defined as at least 45 years of age and 1 year since last regular menses).
17. Participant had a negative urine test result for selected substances of abuse (including alcohol and cotinine) at Screening and Check-in (Day -1).
18. Participant had clinical chemistry, hematology, and complete urinalysis (fasted for at least 8 hours) results within the reference range for the testing laboratory (except results associated with T2DM) unless the out-of-range results were deemed not clinically meaningful by the investigator or sponsor.
19. Participant had a negative test result for hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (anti-HCV), and no known history of human immunodeficiency virus.

Exclusion Criteria:

1. Participant was currently participating in another investigational study or took an investigational drug within 30 days prior to Day 1.
2. Participant received alogliptin previously.
3. Participant was a study site employee, or was an immediate family member (ie, spouse, parent, child, or sibling) of a study site employee involved in conduct of this study.
4. Participant received or donated blood or blood products within 30 days prior to Screening or planned to donate blood during the study.
5. Participant had a known hypersensitivity to alogliptin or related compounds.
6. Participant had a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as consumption of more than 4 alcoholic drinks per day) within 1 year prior to study Day 1.
7. Participant had an acute, clinically significant illness (excluding T2DM) within 30 days prior to study Day 1.
8. Participant had any other condition or prior therapy that, in the opinion of the investigator, would have made the participant unsuitable for the study.
9. Participant had a history or clinical manifestations of significant metabolic (excluding T2DM), hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urologic, immunologic, musculoskeletal, or psychiatric disorder.
10. Participant had a hemoglobin value < 12 g/dL.
11. Participant had a systolic blood pressure > 140 mm Hg or had a diastolic blood pressure > 90 mmHg at Screening or Check-in (Day -1).
12. Adult participant had an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level greater than 2 times the upper limit of normal (ULN), active liver disease, or jaundice at the Screening Visit or on Check-in (Day -1).
13. Pediatric participant had an ALT or AST level greater than 1.5 times the ULN at the Screening Visit or on Check-in (Day -1).
14. Participant had a serum creatinine level > 1.5 mg/dL.
15. Participant had a creatinine clearance (CrCl) < 50 mL/min (normalized to body surface area of 1.73 m^2).
16. Participant had a history of abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy) or thoracic or nonperipheral vascular surgery within 6 months prior to Day 1.
17. Participant had a history or presence of a clinically significant abnormal 12-lead electrocardiogram (ECG) result as determined by the investigator or Takeda at Screening or Check-in (Day -1).
18. Participant had a history of cancer, other than basal cell carcinoma or Stage I squamous cell carcinoma of the skin that had not been in remission for at least 5 years prior to the first dose of study drug.
19. If female, participant was pregnant or lactating or intending to become pregnant before, during, or within 30 days after receiving study drug.
20. If male, participant intended to impregnate others during the study or for 30 days after receiving study drug.
21. Participant consumed or was unable to abstain from consumption of products containing alcohol, caffeine, or xanthine, and food or beverages containing grapefruit juice or Seville-type oranges within 72 hours prior to study Day 1 and for the duration of the study.
22. Participant used any tobacco (ie, nicotine) products (including but not limited to cigarettes, pipe, cigar, chewing tobacco, nicotine patch, or nicotine gum) within 6 weeks prior to study Day 1, and was unwilling to abstain from these products for the duration of the study.
23. Participant used any nutraceutical preparations within 28 days prior to study Day 1.
24. Participant was currently taking ketoconazole, fluconazole, gemfibrozil, rifampin, or carbamazepine or taken within 28 days prior to Check-in (Day -1).
25. Participant had poor peripheral venous access.
26. Participant had a medical history of clinical or laboratory evidence to indicate a diagnosis of type 1 diabetes or secondary forms of diabetes, including maturity-onset diabetes of the young (MODY).

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (7):
- United States (7):
  - Miami, Florida
  - Pineallas Park, Florida
  - Louisville, Kentucky
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States from 17 Sep 2009 to 22 Nov 2013.
Pre-assignment Details: Participants aged 10 to 65 with a diagnosis of type 2 diabetes mellitus were enrolled in 1 of 5 treatment groups and received 12.5 or 25 mg alogliptin once.
Groups:
- Alogliptin 12.5 mg (Age 10 to < 14 Years); Alogliptin 12.5 mg (Age 14 to < 18 Years): Alogliptin 12.5 mg QD, tablets, orally, 1 dose only.
- Alogliptin 25 mg (Age 10 to < 14 Years); Alogliptin 25 mg (Age 14 to < 18 Years); Alogliptin 25 mg (Age 18 to 65 Years): Alogliptin 25 mg QD, tablets, orally, 1 dose only.
Period: Overall Study
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Started | 5 | 4 | 8 | 7 | 22
Completed | 5 | 4 | 7 | 7 | 22
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years) | Total
Number analyzed (Participants) | 5 | 4 | 8 | 7 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (0.89) | 12.0 (0.82) | 15.4 (0.92) | 15.1 (0.69) | 51.3 (8.24) | 31.96 (19.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 5 | 16 | 34
  Male | 1 | 1 | 2 | 2 | 6 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 4 | 7
  Non-Hispanic or Latino | 5 | 3 | 7 | 6 | 18 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  Asian Black or African American | 5 | 3 | 4 | 5 | 15 | 32
  White | 0 | 1 | 4 | 2 | 7 | 14
Height [Mean (Standard Deviation); unit: cm] | 162.4 (8.56) | 165.8 (8.88) | 168.6 (5.71) | 168.9 (9.03) | 167.5 (9.81) | 167.2 (8.73)
Weight [Mean (Standard Deviation); unit: kg] | 86.62 (13.979) | 98.90 (11.957) | 116.28 (33.163) | 103.71 (17.103) | 92.25 (16.454) | 97.14 (21.409)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.22 (4.621) | 36.16 (3.422) | 40.92 (9.190) | 36.46 (6.764) | 32.84 (4.490) | 35.01 (6.439)
Smoking Status [Number; unit: participants]
  Never Smoked | 5 | 4 | 8 | 7 | 14 | 38
  Current Smoker | 0 | 0 | 0 | 0 | 0 | 0
  Ex-smoker | 0 | 0 | 0 | 0 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Alogliptin
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: 1 hour pre-dose and 1, 2, 4, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: Pharmacokinetic set: All participants who received at least 1 dose of study drug and who had at least 1 measureable plasma concentration of alogliptin.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 22
ng/mL | 57.82 (31.5546) | 101.38 (23.4277) | 44.24 (16.7907) | 96.74 (28.3818) | 136.50 (34.2169)

2. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Alogliptin
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: 1 hour pre-dose and 1, 2, 4, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 22
hr | 3.24 (1.1060) | 2.04 (0.0462) | 5.58 (8.2052) | 2.86 (1.4707) | 2.09 (1.1566)

3. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Alogliptin
Description: AUC(0-inf) is measure of area under the curve over the dosing interval (tau) (AUC(0-tau]), where tau is the length of the dosing interval in this study).
Time Frame: 1 hour pre-dose and 1, 2, 4, 8, 12, 16, 24, 48, and 72 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 22
ng•hr/mL | 789.29 (144.0995) | 1221.98 (128.0268) | 688.63 (188.7887) | 1318.41 (123.6279) | 1704.02 (270.6604)

4. Secondary Outcome: Area Under the Plasma Effect-Time Curve From Time 0 to 24 Hours Post-dose (AUEC[0-24]) of Dipeptidyl Peptidase-4 (DPP-4) Inhibition
Description: The area under the plasma effect-time curve from time 0 to 24 hours post-dose (AUEC[0-24]) of dipeptidyl peptidase-4 (DPP-4) inhibition was determined from the inhibition-time curve.
Time Frame: 1 hour pre-dose and 2, 4, 8, 12, and 24 hours post-dose
Population: Pharmacodynamic set: All participants who received at least 1 dose of study drug and who had at least 1 measureable DPP-4 inhibition or GLP-1 concentration.
Measure: Mean (Standard Deviation); unit: Percentage inhibition•hr
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 22
Percentage inhibition•hr | 1569.633 (115.9662) | 1698.852 (74.1622) | 1557.788 (179.5170) | 1854.391 (63.7486) | 1890.012 (71.4549)

5. Secondary Outcome: Maximum Observed Effect (Emax) of Dipeptidyl Peptidase-4 (DPP-4) Inhibition
Description: The maximum observed effect (Emax) of dipeptidyl peptidase-4 (DPP-4) inhibition was determined from the inhibition-time curve.
Time Frame: 1 hour pre-dose and 2, 4, 8, 12, and 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage inhibition
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 22
Percentage inhibition | 83.660 (4.1446) | 89.300 (2.6420) | 81.643 (5.9267) | 90.429 (1.7327) | 92.650 (2.0068)

6. Secondary Outcome: Time to Reach the Maximum Observed Effect of Dipeptidyl Peptidase-4 (DPP-4) Inhibition
Description: The time to reach the maximum observed effect of dipeptidyl peptidase-4 (DPP-4) inhibition was determined from the inhibition-time curve.
Time Frame: 1 hour pre-dose and 2, 4, 8, 12, and 24 hours post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hr
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 22
hr | 4.050 [2.00 to 4.08] | 2.080 [2.00 to 4.00] | 4.000 [2.00 to 4.03] | 4.000 [3.97 to 4.12] | 2.000 [2.00 to 4.07]

7. Secondary Outcome: Observed Effect at 24 Hours Post-dose (E24) of Dipeptidyl Peptidase-4 (DPP-4) Inhibition
Description: The observed effect at 24 hours post-dose (E24) of dipeptidyl peptidase-4 (DPP-4) inhibition was determined from the inhibition-time curve.
Time Frame: 1 hour pre-dose and 2, 4, 8, 12, and 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage inhibition
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 21
Percentage inhibition | 52.000 (10.2976) | 57.375 (5.1292) | 55.400 (9.0239) | 70.400 (5.7660) | 72.843 (5.2949)

8. Secondary Outcome: Area Under the Plasma Effect-Time Curve From Time 0 to 24 Hours Post-dose (AUEC[0-24]) of the Baseline-corrected Glucagon-like Peptide-1 (GLP-1) Concentration
Description: The area under the plasma effect-time curve from time 0 to 24 hours post-dose (AUEC[0-24]) of baseline-corrected glucagon-like peptide-1 was determined from the concentration-time curve. Baseline-corrected glucagon-like peptide-1 concentrations were calculated as the post-dose concentration at each post-dose time point minus the baseline (pre-dose) concentration.
Time Frame: 1 hour pre-dose and 2, 4, 8, 12, and 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol•hr/L
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 21
pmol•hr/L | 117.842 (92.8964) | 120.055 (60.6825) | 168.099 (116.2830) | 122.948 (98.3822) | 278.669 (102.3304)

9. Secondary Outcome: Maximum Observed Effect (Emax) of the Baseline-corrected Glucagon-like Peptide-1 (GLP-1) Concentration
Description: The maximum observed effect (Emax) of baseline-corrected glucagon-like peptide-1 was determined from the concentration-time curve. Baseline-corrected glucagon-like peptide-1 concentrations were calculated as the post-dose concentration at each post-dose time point minus the baseline (pre-dose) concentration.
Time Frame: 1 hour pre-dose and 2, 4, 8, 12, and 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 21
pmol/L | 11.700 (4.6357) | 7.475 (3.8767) | 16.500 (15.0423) | 9.129 (6.6668) | 23.843 (12.1143)

10. Secondary Outcome: Time to Reach the Maximum Observed Effect of the Baseline-corrected Glucagon-like Peptide-1 (GLP-1) Concentration
Description: The time to reach the maximum observed effect of baseline-corrected glucagon-like peptide-1 was determined from the concentration-time curve. Baseline-corrected glucagon-like peptide-1 concentrations were calculated as the post-dose concentration at each post-dose time point minus the baseline (pre-dose) concentration.
Time Frame: 1 hour pre-dose and 2, 4, 8, 12, and 24 hours post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hr
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 21
hr | 8.170 [8.03 to 12.00] | 11.985 [8.00 to 12.00] | 11.920 [8.00 to 12.00] | 8.020 [4.00 to 24.00] | 12.000 [2.33 to 24.02]

11. Secondary Outcome: Observed Effect at 24 Hours Post-dose (E24) of the Baseline-corrected Glucagon-like Peptide-1 (GLP-1) Concentration
Description: The observed effect at 24 hours post-dose (E24) of baseline-corrected glucagon-like peptide-1 was determined from the concentration-time curve. Baseline-corrected glucagon-like peptide-1 concentrations were calculated as the post-dose concentration at each post-dose time point minus the baseline (pre-dose) concentration.
Time Frame: 1 hour pre-dose and 2, 4, 8, 12, and 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Number analyzed (Participants) | 5 | 4 | 7 | 7 | 21
pmol/L | 2.500 (5.3282) | 4.575 (3.6372) | 4.214 (5.2737) | 4.329 (6.2203) | 5.419 (6.2064)

ADVERSE EVENTS:
Description: Safety set: All enrolled participants who received at least 1 dose of study drug.
  At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 12.5 mg (Age 10 to < 14 Years) | Alogliptin 25 mg (Age 10 to < 14 Years) | Alogliptin 12.5 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 14 to < 18 Years) | Alogliptin 25 mg (Age 18 to 65 Years)
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/8 | 0/7 | 0/22
Other Adverse Events (participants affected / at risk) | 3/5 | 1/4 | 5/8 | 2/7 | 9/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg (Age 10 to < 14 Years) (N=5) | Alogliptin 25 mg (Age 10 to < 14 Years) (N=4) | Alogliptin 12.5 mg (Age 14 to < 18 Years) (N=8) | Alogliptin 25 mg (Age 14 to < 18 Years) (N=7) | Alogliptin 25 mg (Age 18 to 65 Years) (N=22)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 4
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 1
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers, nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data, or insights therefrom or any data, information, or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.